CLINICAL TRIAL: NCT01012362
Title: Phase I Study of Pazopanib and Ixabepilone in Patients With Solid Tumors
Brief Title: Study of Pazopanib and Ixabepilone in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS001; 0906M68402 (Other: Institutional Review Board, University of Minnesota); NCI-2009-01444 (Registry Identifier: National Cancer Institute website)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer; Lung Cancer; Colon Cancer; Pancreatic Cancer; Head and Neck Cancer; Kidney Cancer; Sarcoma; Hepatocellular Cancer
Keywords: Solid tumor malignancy; breast cancer; lung cancer; colon cancer; pancreatic cancer; head and neck cancer; kidney cancer; sarcoma; hepatocellular cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Sarcoma; Liver Neoplasms | interventions — pazopanib; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimum Tolerated Dose Determination (Experimental): Patient receives assigned dose level:
  Dose Level 1 = 400 milligrams (mg) of pazopanib and ixabepilone 32 mg/m2. Dose Level 2 = 400 milligrams (mg) of pazopanib and ixabepilone 40 mg/m2. Dose Level 3 = 600 milligrams (mg) of pazopanib and ixabepilone 32 mg/m2. Dose Level 4 = 800 milligrams (mg) of pazopanib and ixabepilone 32 mg/m2.
  Interventions: Drug: Pazopanib; Drug: Ixabepilone
- Optimum Tolerated Dose Confirmation (Experimental): Dose Level 3 = 600 milligrams (mg) of pazopanib and ixabepilone 32 mg/m2.
  Interventions: Drug: Pazopanib; Drug: Ixabepilone

INTERVENTIONS:
Drug: Pazopanib — Escalating doses 400-800 mg by mouth once daily beginning day 1 and continuing.
  Other Names: Pazopanib hydrochloride; GW786034B
Drug: Ixabepilone — Escalating doses 25-32 mg/m2 by intravenous infusion on day 1 of each 21 day cycle
  Other Names: IXEMPRA(TM)

SUMMARY:
This is a Phase I study; dose escalating the combination of pazopanib when taken daily and ixabepilone when administered on day 1 of a 3 week treatment course.

DETAILED DESCRIPTION:
Treatment with ixabepilone will be given at an assigned dose as a 3 hour intravenous infusion on day 1 of a 21 day cycle. Treatment with pazopanib will be given at an assigned dose by mouth once a day, beginning on day 1 and continuing daily. Disease assessment will be done every 2 cycles (6 weeks) with treatment continuing until disease progression, unacceptable toxicity or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced non-hematologic solid tumor malignancy, including, but not limited to breast, lung, colon, pancreatic, head and neck, kidney or sarcoma that has failed or become intolerant to standard therapy and is no longer likely to respond to such therapy Effective with the August 2011 version of the protocol, enrollment is limited to squamous cell carcinoma of the head and neck (refer to section 1.4 for rationale). Note: Patients with a primary diagnosis of hepatocellular carcinoma will be eligible for enrollment into dose level 1 or 2 only, provided they met all other inclusion/exclusion criteria - the maximum tolerated dose (MTD) for pazopanib monotherapy in patients with hepatocellular cancer was found to be 600 mg daily.
* Measureable or evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST).
* Prior systemic chemotherapy, immunotherapy, or biological therapy is allowed; however prior use of either pazopanib or ixabepilone alone or in combination is not allowed.
* At least 14 days must have elapsed since 1) previous systemic therapy (28 days for bevacizumab) before the 1st dose of study drug, 2) last dose of radiation therapy or surgery (28 days for major surgery).
* Patient must have recovered from the acute toxic effects of previous anti-cancer treatment prior to study enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate organ function within 14 days of enrollment defined as:

  * Absolute neutrophil count (ANC) >1.5 x 10^9/L
  * Hemoglobin > or = 9 g/dL
  * Platelets > or = 100 x 10^9/L
  * Prothrombin time or international normalized ratio, and partial thromboplastin time (PTT) < or = 1.2 x upper limit of normal (ULN)
  * Total bilirubin < or = ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < or = 2.5 x ULN
  * Serum creatinine < or = 1.5 mg/dL
  * Urine protein to Creatinine Ratio < 1
  * Total serum calcium < 12.0 mg/dL
* Men and women with child-bearing potential must adhere to protocol criteria to prevent conception during study

Exclusion Criteria:

* Women who are pregnant or nursing.
* Prior radiation to > =or = 30% of major bone marrow containing areas (pelvis, lumbar spine)
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis
* Clinically significant gastrointestinal abnormalities that may increase the risk of GI bleeding or may affect absorption of investigational product
* History of another malignancy - must be at least 3 years disease-free
* Presence of uncontrolled infection
* Prolongation of corrected QT interval (QTc) > 480 msecs
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension
* History of cerebrovascular accident,pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Prior major surgery or trauma within 28 days prior to 1st dose of study drug
* Evidence of active bleeding or bleeding diathesis
* Known endobronchial lesions or involvement of large pulmonary vessels by tumor
* Hemoptysis with 6 weeks of 1st dose of study drug
* Neuropathy Grade 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkaduisz Z Dudek, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Dose Level 1: Pazopanib 400mg - Ixabepilone 32mg/m2
- Arm 1: Dose Level 2: Pazopanib 400mg - Ixabepilone 40mg/m2
- Arm 1: Dose Level 3: Pazopanib 600mg - Ixabepilone 32 mg/m2
- Arm 1: Dose Level 4: Pazopanib 800mg - Ixabepilone 32 mg//m2
- Arm 2: Pazopanib 600mg - Ixabepilone 32 mg/m2. This is an additional cohort of head and neck cancer patients treated at the optimal tolerated regimen for the purpose of performing pharmacokinetics, confirm safety information and obtainadditional preliminary efficacy data in this patient population.
Period: Overall Study
Arm/Group | Arm 1: Dose Level 1 | Arm 1: Dose Level 2 | Arm 1: Dose Level 3 | Arm 1: Dose Level 4 | Arm 2
Started | 9 | 6 | 3 | 4 | 9
Completed | 9 | 6 | 3 | 4 | 9
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Dose Level 1 | Arm 1: Dose Level 2 | Arm 1: Dose Level 3 | Arm 1: Dose Level 4 | Arm 2 | Total
Number analyzed (Participants) | 9 | 6 | 3 | 4 | 9 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 3 | 3 | 7 | 24
  >=65 years | 3 | 1 | 0 | 1 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 1 | 1 | 2 | 11
  Male | 3 | 5 | 2 | 3 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Optimal Tolerated Regimen of Pazopanib and Ixabepilone When Used in Combination
Description: The optimal tolerated regimen is the regimen where ≤ 1 out of 6 patients experiences a dose limiting toxicity (DLT). DLT is defined as one of the following events occurring during cycle 1: grade 4 or greater treatment related hematologic toxicity for > 7 days during the first cycle (21 days) of therapy; grade 3 or greater treatment related clinical non-hematological toxicity (excluding ≥ grade 3 nausea, vomiting, or diarrhea without maximal medical intervention and/or prophylaxis) during the first cycle (21 days) of therapy; or a delay of cycle 2 treatment start by more than 2 weeks due to incomplete hematologic recovery (ANC > 1.5 x 109/L or platelets 100 x 109/L) or unresolved treatment related grade 3 or greater non-hematologic toxicity.
Time Frame: Week 3 of each dose level
Measure: Number; unit: Dose Level
Groups:
- All Arm 1 Participants: All participants who received at least one cycle of one of the following 4 dose levels: Dose Level 1: Pazopanib 400mg - Ixabepilone 32mg/m2; Dose Level 2: Pazopanib 400mg - Ixabepilone 40mg/m2; Dose Level 3: Pazopanib 600mg - Ixabepilone 32 mg/m2; or Dose Level 4: Pazopanib 800mg - Ixabepilone 32 mg//m2.
Arm/Group | All Arm 1 Participants
Number analyzed (Participants) | 22
Dose Level | 3

2. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: A DLT was defined as one of the following events occurring during cycle 1: (1) grade 4 or greater treatment-related hematologic toxicity for >7 days; (2) grade 3 or greater treatment-related clinical non-hematologic toxicity (excluding >/= grade 3 nausea, vomiting, or diarrhea without maximal medical intervention and/or prophylaxis); or (3) delay of starting cycle 2 treatment by >2 weeks due to incomplete hematologic recovery (absolute neutrophil count > 1.5 X 10^9/L or platelets >100 X 10^9/L) or unresolved treatment-related grade 3 or greater non-hematologic toxicity. Adverse events were classified according to Common Terminology Criteria for Adverse Events V 3.0 (CTCAE).
Time Frame: Week 3 of each dose
Population: 6 participants were included at Dose Level 1 to confirm safety after escalation to Dose level 2, but are grouped with the original 3 participants enrolled at Dose Level 1.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Dose Level 1: 400 milligrams (mg) of pazopanib and ixabepilone 32 mg/m2.
- Arm 1: Dose Level 2: 400 milligrams (mg) of Pazopanib and Ixabepilone 40 mg/m2
- Arm 1: Dose Level 3: 600 milligrams (mg) of Pazopanib and Ixabepilone 32 mg/m2
- Arm 1: Dose Level 4: 800 milligrams (mg) of Pazopanib and Ixabepilone 32 mg/m2
- Arm 2: Dose Level 3: 6400 milligrams (mg) of Pazopanib and Ixabepilone 32 mg/m2
Arm/Group | Arm 1: Dose Level 1 | Arm 1: Dose Level 2 | Arm 1: Dose Level 3 | Arm 1: Dose Level 4 | Arm 2: Dose Level 3
Number analyzed (Participants) | 9 | 6 | 3 | 4 | 9
Participants | 0 | 3 | 0 | 1 | 2

3. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: Includes all treatment-related adverse events experienced during and subsequent to Cycle 1.
Time Frame: Up to 30 days post treatment
Population: Dose Level 3 includes participants from Arm 1: Dose Level 3 and Arm 2 combined.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Pazopanib 400mg - Ixabepilone 32mg/m2
- Dose Level 2: Pazopanib 400mg - Ixabepilone 40mg/m2
- Dose Level 3: Pazopanib 600mg - Ixabepilone 32 mg/m2
- Dose Level 4: Pazopanib 800mg - Ixabepilone 32 mg//m2
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 9 | 6 | 12 | 4
Participants | 9 | 6 | 12 | 4

ADVERSE EVENTS:
Groups:
- Dose Level 3: Pazopanib 600mg - Ixabepilone 32 mg/m2 Dose Level 3 includes participants from Arm 1: Dose Level 3 and Arm 2 combined.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Serious Adverse Events (participants affected / at risk) | 4/9 | 3/6 | 7/12 | 3/4
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6 | 12/12 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=9) | Dose Level 2 (N=6) | Dose Level 3 (N=12) | Dose Level 4 (N=4)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 3 | 0
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Decreased Platelets (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Death due to Disease Progression (General disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Chest Wall Pain (General disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Obstruction of Airway (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=9) | Dose Level 2 (N=6) | Dose Level 3 (N=12) | Dose Level 4 (N=4)
Abdominal Bloating (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 6 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 1
Ankle Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 3 | 5 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Bilateral Leg Cramping (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bleeding Gums (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bleeding Neck Wound (General disorders) | 0 | 0 | 1 | 0
Blurred Vision (Eye disorders) | 0 | 0 | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Burning Sensation, Hand (Nervous system disorders) | 0 | 0 | 1 | 0
Chest/Rib Pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1
Decrease Platelets (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Delayed Wound Healing (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 6 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Ear/Head (General disorders) | 0 | 0 | 1 | 0
Edema, Glans Penis (Vascular disorders) | 0 | 0 | 0 | 1
Edema, Limbs (Vascular disorders) | 0 | 0 | 2 | 1
Edema, Periorbital (Eye disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erythema, Arm (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eye Pain (Eye disorders) | 0 | 0 | 1 | 0
Eye Twitch (Eye disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 4 | 4 | 10 | 3
Fever (General disorders) | 0 | 0 | 1 | 0
Fever with Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Flu-Like Syndrome (General disorders) | 0 | 0 | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Folliculitis, Leg (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Fracture, Arm (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fungal Infection, Feet (Infections and infestations) | 0 | 0 | 1 | 0
Genreralized Body Aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hand Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 4 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hemoglobin, NOS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypopigmentation, Eyelashes and Eyebrows (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypopigmentation, Hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Increased Liver Enzyme, ALT (Investigations) | 0 | 0 | 0 | 1
Increased Liver Enzyme, AST (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Increased Sweating (General disorders) | 0 | 0 | 1 | 0
Increased Trachea Secretions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Infection, Lung (Infections and infestations) | 0 | 0 | 1 | 0
Infection, NOS (Infections and infestations) | 0 | 0 | 1 | 0
Infection, Port Incision (Infections and infestations) | 0 | 0 | 1 | 0
Infection, Urinary (Infections and infestations) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Jaw/Neck Wound Pain (General disorders) | 0 | 0 | 1 | 0
Joint Pain (General disorders) | 1 | 1 | 4 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Leg Pain (General disorders) | 0 | 0 | 0 | 1
Leukocytes, NOS (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Leukocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphedema (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Mucositis (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 9 | 2
Neck Pain (General disorders) | 1 | 0 | 0 | 0
Neuropathy, NOS (Nervous system disorders) | 1 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 6 | 4 | 1
Neutrophils, NOS (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 (0)
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Partial Thromboplastin Time, NOS (Investigations) | 0 | 0 | 1 | 0
Peripheral Neuropathy (Nervous system disorders) | 0 | 0 | 4 | 1
Platelets, NOS (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 0
Reflux (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinnorhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Scrotal Cysts (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Sinus Infection (Infections and infestations) | 0 | 0 | 1 | 1
Skin Breakdown near Gastrostomy Tube (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Stomach Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Taste Alteration (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Throat Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Leakage (Renal and urinary disorders) | 1 | 0 | 0 | 0
Viral Infection, NOS (Infections and infestations) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 6 | 2
Weakness, NOS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Weepy Scalp (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Weight Loss (Investigations) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No